CLINICAL TRIAL: NCT04467112
Title: Non Inferiority Trial for Detection of nCOVID-19 Through Analysis of Exhaled Breath Aerosols
Status: Completed | Type: Observational
Sponsor: Owlstone Ltd (Industry)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-Breath
Record Dates: First submitted 2020-06-30; First posted 2020-07-10 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The face mask will be placed onto the subject's face, covering his/her nose and mouth, head straps will be used to ensure that the face mask is kept in place for the duration of the test. This mask will contain a material designed to capture exhaled respiratory droplets and/or aerosols. Several iterations of these impaction and filtration devices may be used to optimize functional attributes of the material for capture of COVID. These materials will always have a proven safety for use with humans.
  Subjects can talk, cough and sneeze in the mask or can temporarily remove the mask if uncomfortable, to drink some water etc if required. Total collection time spread across two masks will not exceed one hour
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Breath Biopsy face masks with removable filters and fitted PVA strip — Device developed for collection of breath samples

SUMMARY:
This study aims to evaluate several of Owlstone Medical's Breath Biopsy aerosol respiratory droplet capture techniques for the detection of nCOVID-19.

These are single use disposable breath capture devices with removable filters and fitted PVA strip that directly sample exhaled breath aerosols and therefore, directly sample the primary transmission route for the virus. They can be used independently and shipped for analysis for the presence of nCOVID-19 using established existing assays available in any reference lab.

The trial is a non-inferiority trial comparing diagnostic accuracy of collection via face mask vs. available diagnostic procedures in standard care and will also asses the feasibility of patient use of the equipment.

Subjects will be recruited at the Addenbrookes Hospital, Cambridge. Minimal patient characteristics (e.g. age, sex) are collected.

Between 20 and 100 subjects with with a positive nCOVID-19 diagnosis will be sampled to obtain to address the primary study hypothesis. Due to the pre-test probability of patients being positive for nCOVID-19 is unknown we will monitor the number of sampled subjects with a positive diagnosis on a weekly basis. The clinical diagnosis of the subject based on a combination of imaging, viral diagnostics and clinical assessment will be used as the reference standard. When this number hits 100 the study will be discontinued. In total no more than 500 subjects shall be sampled in this trial.

DETAILED DESCRIPTION:
Subjects will be recruited for the study during their scheduled appointments per clinical practice to the site, no separate study visit is required.

The participant's involvement in the study will be limited to one visit (per routine practice) only. No additional follow up is required.

For the purpose of the study a breath sample will be collected using the Breath Biopsy face masks. Collection of exhaled breath aerosols using these single use, disposable face masks will require subjects to breath normally into these face masks, the total collection time will not exceed one hour. It is expected to reduce collection times after initial validation steps to the shortest time providing sufficient diagnostic accuracy.

Given the non-invasive nature of these breath collections subjects can immediately provide up to two samples using the Breath Biopsy face masks. The breath collection should occur within 24 hours of the diagnostic sample.

Collected samples will be either frozen or shipped for rtPCR analysis of the presence of nCOVID-19 RNA. The two Breath Biopsy face masks can be used as technical replicates and/or to validate different storage conditions.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Be 16 years or older
* Suspected or confirmed nCOVID-19 infection

Exclusion Criteria:

* Subjects unable to provide written informed consent
* Ineligible subjects will specifically include subjects:

  * deemed unlikely to be able to maintain oxygen saturation of greater than 90% while breathing room air for 30 seconds Require non-invasive ventilation or high flow nasal oxygen
  * who require inotropic medication to maintain adequate organ perfusion
  * communication barrier and / or unable to comply with the instructions to use the Breath Biopsy face masks

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The inclusion and exclusion criteria for the various study populations are detailed above. General inclusion and exclusion criteria which apply to all study subjects are detailed followed by indication specific criteria are also detailed for both inclusion and exclusion.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Detection of nCOVID-19 using a face mask | 1 year
  The primary aim of this study is to establish non-inferiority of the Breath Biopsy face masks with various respiratory droplet (aerosol) capture techniques for the detection of nCOVID-19 compared to the current diagnostic test results per standard practice.

SECONDARY OUTCOMES:
Independent Patient use of face mask | 1 year
  The secondary objective is to assess the feasibility of independent use of the Breath Biopsy face masks. This will be measured by means of patient reported feedback on their level of comfort in performing the breath collection

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Marciniak, Study Chair — Cambridge Institute for Medical Research
Locations (1):
- Cambridge University Hospital NHS, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No